CLINICAL TRIAL: NCT03094559
Title: Correlation Between FlowMet™, ABI, SPP, TBI, TcPO2 and Angiography
Brief Title: Correlation Between FlowMet™ and Other Gold Standard Assessments in the Management of Critical Limb Ischemia (CLI)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator leaving institution
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16-1223
Record Dates: First submitted 2017-03-07; First posted 2017-03-29 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Critical Limb Ischemia
Keywords: peripheral arterial disease
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FlowMet device (Experimental): This is a feasibility study
  Interventions: Device: FlowMet

INTERVENTIONS:
Device: FlowMet — The FlowMet device will be placed on the index finger of the right hand. Signal fidelity will be assured by confirming the presence of a pulse waveform if one is expected and by assuring that an appropriate amount of light is be detected by the FlowMet device. Following placement of the FlowMet device, a period of 10 seconds will be allowed to elapse to allow transient changes in perfusion due to device placement to diminish. FlowMet blood flow data will be recorded for 20 seconds using the FlowMet data acquisition software. These steps will be repeated for digits 1 and 2 on the limb with diagnosed or suspected CLI, or on both limbs if both are diagnosed or suspected of having CLI.

SUMMARY:
The purpose of this study is to demonstrate the utility of the FlowMet™ device in the assessment of perfusion in subjects suspected of or being treated for critical limb ischemia, in comparison to other gold standard technologies, such as ankle brachial pulse index (ABI), skin perfusion pressure (SPP), toe brachial pulse index (TBI), transcutaneous oxygen tension (TcP02), and angiography currently in use in the clinic.

DETAILED DESCRIPTION:
TRIAL OBJECTIVES

1.0

To demonstrate that the FlowMet is effective for the assessment of tissue perfusion compared to gold standard technologies in patients suspected of or being treated for CLI.

2.0 STUDY DESIGN

This is a single center, cross-sectional study of subjects who are scheduled for CLI assessment with a Rutherford score of V and VI.

The subjects will be evaluated at baseline for determination if they meet the inclusion/exclusion criteria of the protocol. If the subject is eligible to enroll in the trial and they have signed an informed consent form (ICF) and are scheduled for evaluation, they will be enrolled. Subjects will undergo FlowMet, ABI, SPP, TBI, TcPO2, and angiography measurements (if not performed previously). The correlation between the aforementioned standard clinical measurements and FlowMet measurements will be assessed.

As ABI, SPP, TBI, TcPO2, Rutherford score, time of surgical (re)admission, speed of wound healing, and angiography measurements will likely change over a period of one year following initial FlowMet measurements, future measurements up to one year post FlowMet measurement (and performed as a standard of care) may also be correlated to initial FlowMet measurements to assess the whether FlowMet data is correlated to long-term patient outcomes.

3.0 STUDY PROCEDURES

3.1 Randomization, Blinding and Subject Identification

This is a cross-sectional study of subjects being treated for CLI with a Rutherford score of V or VI. No randomization scheme is required.

3.2 Product Equipment (FlowMet)

All parts of the FlowMet were manufactured in facilities with ISO 9001:2008 certification. Instruments are constructed in an ISO 9 cleanroom. All materials intended to be in contact with the patient's skin are constructed of polydimethylsiloxane (silicone) rubber which was sterilized via autoclave prior to device construction. Polydimethylsiloxane is widely used in existing medical devices and has been shown to be safe for both short-term contact, as well as long-term implantation (The AMS Sphincter 800™ Urinary Prosthesis, PMA P000053). Between uses, all polydimethylsiloxane components, in addition to all components which can accidentally contact a patient's skin during use, can be sanitized using alcohol wipes or germicidal wipes, such as alcohoPSI Inc. Sani-Cloths, which are commonly used in hospitals and which are bactericidal, tuberculocidal, and virucidal. The FlowMet has been used on 37 patients without adverse events at the University of California, Irvine in a study of tissue optical properties approved and overseen by the University of California, Irvine IRB. The FlowMet has not been evaluated, cleared or approved for use by the FDA.

3.3 Details of FlowMet usage

Extremity perfusion measurements will be performed using the FlowMet peripheral perfusion device. All extremity blood flow measurements will be collected during room air inhalation.

3.3.1

i. The FlowMet device will be placed on the index finger of the right hand. Signal fidelity will be assured by confirming the presence of a pulse waveform if one is expected and by assuring that an appropriate amount of light is be detected by the FlowMet device. The following light intensity values are acceptable: maximum intensity greater than 25 but less than 255 and average subtracted intensity greater than 20 but less than 175.

ii. Following placement of the FlowMet device, a period of 10 seconds will be allowed to elapse to allow transient changes in perfusion due to device placement to diminish.

iii. FlowMet blood flow data will be recorded for 20 seconds using the FlowMet data acquisition software.

iv. Steps i-iii will be repeated for digits 1 and 2 on the limb with diagnosed or suspected CLI, or on both limbs if both are diagnosed or suspected of having CLI. All data sets will be saved, and blood flow in each digit will be computed as the average of the collected data over the 20 second data collection period. If alternative digits are used for data acquisition due to differences in physiology, this will be recorded. If subject is missing the aforementioned toes, the tester will choose a different set of digits and this change will be recorded.

4.0 STUDY PROCEDURES

4.1 Baseline and Assessment

The Cleveland Clinic's standard of care will be followed for all participating study subjects. The following procedures will be conducted as part of a baseline assessment:

* Informed consent
* Complete medical history
* Demographics
* Vital signs (heart rate and blood pressure), height and weight
* Record angiographic data for study (if available)

The following procedures are standard of care and will be conducted to assess perfusion:

* Ankle brachial pulse index (ABI)
* Skin Perfusion Pressure (SPP)
* Toe brachial pulse index (TBI)
* Transcutaneous oxygen tension (TcP02)
* Angiography (if not performed previously)

The following procedures are not standard of care and will be conducted to assess perfusion:

* FlowMet measurement on subject's hand and foot/feet

ELIGIBILITY:
Inclusion Criteria:

* Subject is willing and able to provide an informed consent.
* Subject is willing and able to comply with the study procedures.
* Subject is able to understand the study procedures.
* Subject is being seen at the clinic for the evaluation/treatment of CLI.
* Subject has a Rutherford score of V or VI.

Exclusion Criteria:

* Subject has any medical condition, which in the judgment of the Investigator and/or designee makes the subject a poor candidate for the investigational procedure
* Anyone with a latex allergy
* Must be over 18 years old
* Must not be pregnant during time of study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-03-07 (Actual); Primary Completion 2018-01 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Correlation between FlowMet perfusion values and ankle-brachial index and toe-brachial index in 34 patients who present to outpatient clinic. | One year
  Correlation between FlowMet perfusion values evaluating the median systolic, median diastolic, and overall flow and amplitude as compared to ABI and TBI. This is a feasibility study to determine the degree of correlation between this novel device and current standard of care testing to see how the numerical values obtained correlate with both normal and abnormal values of well established testing. Normal values of ABI (ratios of > 0.9 to < 1.3) and TBI (ratios of > 0.7).
Correlation between FlowMet perfusion values and skin perfusion pressure in 34 patients who present to outpatient clinic. | One year
  Correlation between FlowMet perfusion values evaluating the median systolic, median diastolic, and overall flow and amplitude as compared to skin perfusion pressure testing. This is a feasibility study to determine the degree of correlation between this novel device and current standard of care testing to see how the numerical values obtained correlate with both normal and abnormal values of well established testing. Normal values of SPP are 40-50 mmHg.
Correlation between FlowMet perfusion values and transcutaneous oxygen tension in 34 patients who present to outpatient clinic. | One year
  Correlation between FlowMet perfusion values evaluating the median systolic, median diastolic, and overall flow and amplitude as compared to transcutaneous oxygen testing. This is a feasibility study to determine the degree of correlation between this novel device and current standard of care testing to see how the numerical values obtained correlate with both normal and abnormal values of well established testing. Normal value at the foot is 40-50 mmHg.
Correlation between FlowMet perfusion values and angiography in 34 patients who present to outpatient clinic. | One year
  Correlation between FlowMet perfusion values evaluating the median systolic, median diastolic, and overall flow and amplitude as compared to angiography. This is a feasibility study to determine the degree of correlation between this novel device and current standard of care testing to see how the numerical values obtained correlate with both normal and abnormal angiographic images as defined by severity of stenosis.

SECONDARY OUTCOMES:
Correlation between FlowMet perfusion values and Rutherford score | One year
  Correlation between FlowMet perfusion values evaluating the median systolic, median diastolic, and overall flow and amplitude as compared to Rutherford score of patient at time of evaluation.
Correlation between FlowMet perfusion values and time of surgical (re)admission | One year
  Correlation between FlowMet perfusion values evaluating the median systolic, median diastolic, and overall flow and amplitude to determine timing of surgical (re)admission (days).
Correlation between FlowMet perfusion values and speed of wound healing | One year
  Correlation between FlowMet perfusion values evaluating the median systolic, median diastolic, and overall flow and amplitude to determine speed of wound healing (days).

CONTACTS AND LOCATIONS:
Overall Officials: Mehdi Shishehbor, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD

REFERENCES:
- [Background] Anderson RR, Parrish JA. The optics of human skin. J Invest Dermatol. 1981 Jul;77(1):13-9. doi: 10.1111/1523-1747.ep12479191. PMID 7252245
- [Background] Wilson BC, Adam G. A Monte Carlo model for the absorption and flux distributions of light in tissue. Med Phys. 1983 Nov-Dec;10(6):824-30. doi: 10.1118/1.595361. PMID 6656695
- [Background] Got I. [Transcutaneous oxygen pressure (TcPO2): advantages and limitations]. Diabetes Metab. 1998 Sep;24(4):379-84. French. PMID 9805653
- [Background] Zwicky S, Mahler F, Baumgartner I. Evaluation of clinical tests to assess perfusion in chronic critical limb ischemia. Vasa. 2002 Aug;31(3):173-8. doi: 10.1024/0301-1526.31.3.173. PMID 12236021
- [Background] Jakobsson A, Nilsson GE. Prediction of sampling depth and photon pathlength in laser Doppler flowmetry. Med Biol Eng Comput. 1993 May;31(3):301-7. doi: 10.1007/BF02458050. PMID 8412384
- [Background] Sprengers RW, Teraa M, Moll FL, de Wit GA, van der Graaf Y, Verhaar MC; JUVENTAS Study Group; SMART Study Group. Quality of life in patients with no-option critical limb ischemia underlines the need for new effective treatment. J Vasc Surg. 2010 Oct;52(4):843-9, 849.e1. doi: 10.1016/j.jvs.2010.04.057. PMID 20598482
- [Background] Varu VN, Hogg ME, Kibbe MR. Critical limb ischemia. J Vasc Surg. 2010 Jan;51(1):230-41. doi: 10.1016/j.jvs.2009.08.073. PMID 20117502
- [Background] Hirsch AT, Hartman L, Town RJ, Virnig BA. National health care costs of peripheral arterial disease in the Medicare population. Vasc Med. 2008 Aug;13(3):209-15. doi: 10.1177/1358863X08089277. PMID 18687757
- [Background] Norgren L, Hiatt WR, Dormandy JA, Nehler MR, Harris KA, Fowkes FG; TASC II Working Group; Bell K, Caporusso J, Durand-Zaleski I, Komori K, Lammer J, Liapis C, Novo S, Razavi M, Robbs J, Schaper N, Shigematsu H, Sapoval M, White C, White J, Clement D, Creager M, Jaff M, Mohler E 3rd, Rutherford RB, Sheehan P, Sillesen H, Rosenfield K. Inter-Society Consensus for the Management of Peripheral Arterial Disease (TASC II). Eur J Vasc Endovasc Surg. 2007;33 Suppl 1:S1-75. doi: 10.1016/j.ejvs.2006.09.024. Epub 2006 Nov 29. No abstract available. PMID 17140820
- [Background] Falanga V. Wound healing and its impairment in the diabetic foot. Lancet. 2005 Nov 12;366(9498):1736-43. doi: 10.1016/S0140-6736(05)67700-8. PMID 16291068
- [Background] Ouriel K. Peripheral arterial disease. Lancet. 2001 Oct 13;358(9289):1257-64. doi: 10.1016/S0140-6736(01)06351-6. PMID 11675083
- [Background] Cronberg CN, Sjoberg S, Albrechtsson U, Leander P, Lindh M, Norgren L, Danielsson P, Sonesson B, Larsson EM. Peripheral arterial disease. Contrast-enhanced 3D MR angiography of the lower leg and foot compared with conventional angiography. Acta Radiol. 2003 Jan;44(1):59-66. PMID 12631001
- [Background] Stadelmann WK, Digenis AG, Tobin GR. Impediments to wound healing. Am J Surg. 1998 Aug;176(2A Suppl):39S-47S. doi: 10.1016/s0002-9610(98)00184-6. PMID 9777971
- [Background] Mosely LH, Finseth F. Cigarette smoking: impairment of digital blood flow and wound healing in the hand. Hand. 1977 Jun;9(2):97-101. doi: 10.1016/s0072-968x(77)80001-6. PMID 914099
- [Background] Prahl, S. A., Keijzer, M., Jacques, S. L. & Welch, A. J., SPIE Proceedings of Dosimetry of Laser Radiation in Medicine and Biology. 102-111 (Proc. SPIE IS 5, 1989).
- [Background] Hirsch AT, Haskal ZJ, Hertzer NR, Bakal CW, Creager MA, Halperin JL, Hiratzka LF, Murphy WR, Olin JW, Puschett JB, Rosenfield KA, Sacks D, Stanley JC, Taylor LM Jr, White CJ, White J, White RA, Antman EM, Smith SC Jr, Adams CD, Anderson JL, Faxon DP, Fuster V, Gibbons RJ, Halperin JL, Hiratzka LF, Hunt SA, Jacobs AK, Nishimura R, Ornato JP, Page RL, Riegel B; American Association for Vascular Surgery; Society for Vascular Surgery; Society for Cardiovascular Angiography and Interventions; Society for Vascular Medicine and Biology; Society of Interventional Radiology; ACC/AHA Task Force on Practice Guidelines; American Association of Cardiovascular and Pulmonary Rehabilitation; National Heart, Lung, and Blood Institute; Society for Vascular Nursing; TransAtlantic Inter-Society Consensus; Vascular Disease Foundation. ACC/AHA 2005 guidelines for the management of patients with peripheral arterial disease (lower extremity, renal, mesenteric, and abdominal aortic): executive summary a collaborative report from the American Association for Vascular Surgery/Society for Vascular Surgery, Society for Cardiovascular Angiography and Interventions, Society for Vascular Medicine and Biology, Society of Interventional Radiology, and the ACC/AHA Task Force on Practice Guidelines (Writing Committee to Develop Guidelines for the Management of Patients With Peripheral Arterial Disease) endorsed by the American Association of Cardiovascular and Pulmonary Rehabilitation; National Heart, Lung, and Blood Institute; Society for Vascular Nursing; TransAtlantic Inter-Society Consensus; and Vascular Disease Foundation. J Am Coll Cardiol. 2006 Mar 21;47(6):1239-312. doi: 10.1016/j.jacc.2005.10.009. No abstract available. PMID 16545667